CLINICAL TRIAL: NCT05442164
Title: Effect of Implementation of the Danish Emergency Surgery (DANAKIR) Support Network on Post-discharge Outcomes After Major Emergency Abdominal Surgery: a Prospective Before And-after Study
Brief Title: Effect of Implementation of the Danish Emergency Surgery (DANAKIR) Support Network on Post-discharge Outcomes After Major Emergency Abdominal Surgery
Acronym: DANAKIR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Dunja Kokotovic, Doctor, Postdocteral fellow, Herlev Hospital
Other Study IDs: DANAKIR
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Bowel Perforated; Bowel Obstruction
MeSH Terms: conditions — Intestinal Perforation; Intestinal Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before-group: Patients undergoing major emergency surgery before a supportive network is established
- After-group: Patients undergoing major emergency surgery after a supportive network is established
  Interventions: Behavioral: DANAKIR support network

INTERVENTIONS:
Behavioral: DANAKIR support network — The DANAKIR intervention will consist of:
  * Structured written discharge information
  * Invitation to the DANAKIR monthly information meeting DANAKIR meetings The monthly meetings are a core component of the support network. One time each month, a meeting will be held at Herlev Hospital with the participation of an emergency surgeon, an emergency surgery dedicated nurse, a dietician, and a physiotherapist. Each professional (surgeon, nurse, dietician, physiotherapist) will host an informative 15 minute session regarding the postoperative course after major emergency surgery. Following the presentations time for questions in plenum and private with the different experts will be held. Furthermore, there will be an opportunity for networking at the DANAKIR meeting. Each meeting is planned to last 2 hours. At the end of each meeting the patients will be asked to evaluate the meeting and content.
  Groups: After-group

SUMMARY:
Effect of implementation of the Danish Emergency Surgery (DANAKIR) support Network on post-discharge outcomes after major emergency abdominal surgery: a prospective before and-after study

Background Major emergency abdominal surgery is performed in more than 5000 patients yearly in Denmark. In general, little is known about the period after the discharge of these patients besides that chronic pain, physical dysfunction, and quality of life are severely affected in up to 50% of patients at long-term follow-up. A recent study investigating unplanned readmission after major emergency abdominal surgery found that up to 50% undergo unplanned readmission within the first 180 days after discharge.

Purpose The purpose of this study is to evaluate the effects of inviting patients undergoing major emergency surgery and their relatives to join a support network after discharge (the DANAKIR network).

Methods This study is designed as a before- and after study. Prior to establishing the DANAKIR (Danish Emergency Surgery Network) support network, the investigators will consecutively during a one year inclusion period prospectively include all patients undergoing emergency abdominal surgery with a midline laparotomy. The inclusion period starts 1st August 2021.

The investigators will register the following in the pre-implementation phase:

* Postoperative day (POD) 30: Quality of life (EQ-5D-5L) (by telephone)
* POD90: Quality of life (EQ-5D-5L) (by telephone), readmissions (by hospital file)
* POD 180: Quality of life (EQ-5D-5L) (by telephone), readmissions (by hospital file)
* Number of days at home with 90 days (by hospital file)
* Number of participants with at least one readmission (by hospital file) Hereafter the investigators will establish the DANAKIR support network. The investigators plan for a six-month inclusion period with DANAKIR starting 1th of September 2022

Intervention

The DANAKIR intervention will consist of:

* Structured written discharge information for the participanats and relatives about expectations and precautions
* Invitation to the DANAKIR monthly information meeting All patients undergoing emergency abdominal surgery and members of their family are invited to participate in at least one DANAKIR meeting. Patients and their relatives can participate in as many meetings as they wish; however, we encourage all patients to participate at least once.

DANAKIR meetings The monthly meetings are a core component of the support network. One time each month, a meeting will be held at Herlev Hospital with the participation of an emergency surgeon, an emergency surgery dedicated nurse, a dietician, and a physiotherapist. Furthermore, there will be research personnel present. Each professional (surgeon, nurse, dietician, physiotherapist) will host an informative 15 minute session regarding the postoperative course after major emergency surgery. Following the presentations time for questions in plenum and private with the different experts will be held. Furthermore, there will be an opportunity for networking at the DANAKIR meeting. Each meeting is planned to last 2 hours. At the end of each meeting the patients will be asked to evaluate the meeting and content.

Outcome measures The primary outcome of this study is the number of days at home within 90 days of surgery. The secondary outcomes are quality of life at 30 days, 90 days, and 180 days after surgery and the number of patients with at least one emergency readmission 90 days and 180 days from surgery.

Trial size The investigators expect to include 200 patients in the before group and 200 patients in the after group.

Perspectives The DANAKIR support network examines if a structure with physical network meetings is effective in regard to quality of life and preventing readmissions after major emergency surgery. The investigators hypothesize that the days at home will increase within 90 days from surgery and that quality of life will increase for both participants and their relatives by implementing a simple and obvious solution. If the DANAKIR network proves efficient it is an easily implemented solution to increase quality of life and days at home after major emergency surgery.

ELIGIBILITY:
Inclusion Criteria:

* Emergency open, laparoscopic or laparoscopically assisted procedures involving: stomach, small bowel, large bowel, or rectum for conditions such as perforation, ischemia, abdominal abscess, bleeding, haematoma, or obstruction
* Bowel resection due to incarcerated incisional, umbilical, inguinal, and femoral hernias (but not hernia repair without bowel resection/repair)
* Laparoscopic/open adhesiolysis
* Fascial dehiscence
* Emergency surgery after elective surgery if criteria above is met

Exclusion Criteria:

* Elective procedures
* Appendectomy +/- drainage of localized abscess
* Cholecystectomy +/- drainage of localized abscess
* Emergency hernia repair without bowel resection
* Large-bowel endoscopic stent procedures
* Superficial wound dehiscence above the fascia
* Ruptured ectopic pregnancy or pelvic abscess due to inflammatory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at the department of Surgery, Herlev Hospital. A large University Hospital in the Capital Region of Denmark
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Days at home within 90 days | 90 day
  Number of days at home within 90 days of surgery

SECONDARY OUTCOMES:
Quality of life | Day 30, day 90, day 180
  EQ-5D-5L
Readmission | Day 90 and day 180
  number of patients with at least one emergency readmission

IPD SHARING:
Plan to Share IPD: No